CLINICAL TRIAL: NCT06801366
Title: VIdeo Clips for Diagnostic Evaluation of Obstructive Sleep Apnea in Children (VIDEO)
Brief Title: VIdeo Clips for Diagnostic Evaluation of Obstructive Sleep Apnea in Children
Acronym: VIDEO
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital of Eastern Ontario (Other)
Responsible Party: Principal Investigator, Sherri Katz, Division Chief of Pediatric Respirology and Senior Scientist, Children's Hospital of Eastern Ontario
Other Study IDs: 24/19CTO; 517815 (Other Grant/Funding Number: CIHR)
Record Dates: First submitted 2025-01-24; First posted 2025-01-30 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Obstructive Sleep Apnea (OSA)
Keywords: obstructive sleep apnea; polysomnography; videos
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with suspected Obstructive Sleep Apnea: Children referred for polysomnography (PSG) to investigate symptoms of obstructive sleep apnea (OSA).
  Interventions: Diagnostic Test: Parent-recorded smartphone video clips

INTERVENTIONS:
Diagnostic Test: Parent-recorded smartphone video clips — Parents will record smartphone video clips of their child asleep, which will be scored by pediatric sleep physicians for presence of moderate-severe OSA. Children will then undergo clinically indicated polysomnography (PSG). Video clips will be evaluated for diagnostic accuracy, with PSG as the gold standard.

SUMMARY:
Obstructive sleep apnea (OSA), which occurs in 1-4% of children, is a serious condition where a person stops breathing periodically during sleep because their airway closes. Untreated, it is associated with high blood pressure, behavioural problems, and lower quality of life. While early diagnosis and treatment are critical, there are significant barriers to access to a sleep study (the best diagnostic test). Questionnaires and overnight oxygen level recordings are limited in their ability to identify OSA. Better screening tools are needed to identify and prioritize children for sleep study testing. Short video clips, recorded using smartphones by parents, may be a useful tool to identify children at risk of OSA who would most benefit from a sleep study. The study aims to evaluate the ability of home smartphone video clips as a screening tool for moderate-severe OSA in children referred for a sleep study. The utility of video clips will also be compared to questionnaires and overnight oxygen saturation recordings. The investigators believe that the video clips will be able to predict moderate-severe OSA in children and that they will be better than standard clinical questionnaires or oxygen recordings. This multi-centre study will include 625 children referred for sleep studies for suspected OSA. Parents will be asked to record short video clips of their child sleeping, which will be rated for the presence and severity of OSA. Children will then undergo a sleep study, and parents will complete a questionnaire about sleep symptoms. Oxygen level recordings will be extracted from the sleep study. The diagnostic accuracy of video clips will be determined and compared to the questionnaire and oxygen level recording. This new approach to screening for pediatric OSA using widely available technology will allow children at the highest risk for moderate-severe OSA to be diagnosed and treated earlier, minimizing the risk of long-term complications.

ELIGIBILITY:
Inclusion Criteria:

* 2-18 years old
* referred for diagnostic PSG to assess for OSA at their local tertiary care centre
* parent/caregiver has access to mobile technology

Exclusion Criteria:

* previous diagnosis of sleep-disordered breathing based on PSG in the last five years
* unable to cooperate for PSG
* clinician-suspected presence of central sleep apnea or central hypoventilation
* genetic or congenital syndrome
* non-verbal
* use of PAP therapy or tracheostomy
* parent/caregiver does not speak English or French

Ages: 2 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: 4 Canadian tertiary pediatric centres: Children's Hospital of Eastern Ontario (Ottawa), The Hospital for Sick Children (Toronto), Montreal Children's Hospital (Montreal), Stollery Children's Hospital (Edmonton)
Sampling Method: Non-Probability Sample
Enrollment: 625 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of video clips | From enrolment to end of data analysis (5 years).
  Evaluate the diagnostic accuracy of video clips compared to PSG in the detection of moderate-severe OSA. Estimate the area under the ROC curve.

SECONDARY OUTCOMES:
Specificity of video clips | From enrolment until the end of data analysis (5 years)
  To determine the specificity of video clips for diagnosis of moderate-severe OSA, if sensitivity is held at 0.90.
Sensitivity of video clips | From enrolment until the end of data analysis (5 years)
  To determine the sensitivity of video clips for diagnosis of moderate-severe OSA, if specificity is held at 0.90.
The added benefit of oximetry to the accuracy of video clips | From enrolment until the end of data analysis (5 years)
  To determine the added benefit of oximetry to the specificity and sensitivity of the video clips, if each is individually held at 0.90.
The added benefit of the Pediatric Sleep Questionnaire (PSQ) and oximetry to the accuracy of video clips | From enrolment until the end of data analysis (5 years)
  To further determine the benefit of the PSQ in addition to oximetry and video clips in terms of specificity and sensitivity, if each is individually held at 0.90.

CONTACTS AND LOCATIONS:
Locations (4):
- Canada (4):
  - Stollery Children's Hospital, Edmonton, Alberta
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - Montreal Children's Hospital, Montreal, Quebec